CLINICAL TRIAL: NCT02188940
Title: Effects of Exercise Training in a Weight-loss Lifestyle Intervention on Clinical Control and Psychosocial Morbidity in Obese Asthmatics: a Randomized and Controlled Trial
Brief Title: Exercise Training to Lose Weight in Obese Asthmatics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: University of Sao Paulo (Other); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ETLWOA; 2012/16700-9 (Other Grant/Funding Number: São Paulo Research Foundation (FAPESP))
Record Dates: First submitted 2014-07-10; First posted 2014-07-14 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2014-07

CONDITIONS: Asthma; Obesity
Keywords: Asthma; Obesity; Clinical control; Exercise; Weight-loss
MeSH Terms: conditions — Asthma; Obesity; Motor Activity; Weight Loss | interventions — Diet; Early Intervention, Educational; Behavior Therapy; Exercise; Breathing Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise, dietary and behavioral therapy (Active Comparator): The interventions of active comparator will be education program, dietary and behavioral therapy and exercise training.
  Interventions: Behavioral: Dietary; Behavioral: Education Program; Behavioral: Behavioral Therapy; Other: Exercise Training
- Dietary and behavioral therapy (Sham Comparator): The intervention in sham comparator will be education program, dietary and behavioral therapy and stretching and breathing exercise.
  Interventions: Behavioral: Dietary; Behavioral: Education Program; Behavioral: Behavioral Therapy; Other: Stretching and Breathing exercise

INTERVENTIONS:
Behavioral: Dietary — The dietary therapy will be performed every 15 days, totaling 6 sessions of 60 minutes each by a dietitian. Patients will be advised to follow restricted-calorie diet based on the hypocaloric dietary guidance, multiplying the patient's weight by 20 to 25 calories. The Nutwin ® program will be used to structure the patient's diets, based on 24 hours food record and calories tables. Throughout the program, issues related to food control, the benefits of following a balanced diet and the changing food habits will be discussed.
Behavioral: Education Program — The education program will consist of 4 classes lasting 6 hours at the beginning of the interventions, in which issues related to asthma and physical activity will be discussed. Presentations and group discussions will be carried out, including information about asthma pathophysiology, medication and peakflowmeter skills, self-monitoring techniques, environmental control, benefits and current recommendations of physical activity.
Behavioral: Behavioral Therapy — The Behavioral therapy will be performed every 15 days, totaling 6 sessions of 60 minutes each by a psychologist. Sessions of group dynamics will be performed to increase the patient adherence in a weight loss program using behavior modification techniques, such as self-management, motivational strategies, positive reinforcement and relapse prevention. Relaxation techniques, experiences and patient's report will also be used.
Other: Exercise Training — The aerobic training will be performed on a treadmill and a bike (or an elliptical), twice a week, totaling 24 sessions of 60 minutes each. The initial intensity will be 50% to 60% of VO2 max reaching a maximal 75% of VO2 max and the progression will take place according to the level of effort (Borg) in the last two sessions. Patients will be advised to walk outside at least twice a week for 30 minutes and write down their activity in a diary. Furthermore, they will be given an accelerometer in week 6 to record their daily steps. The resistance training will consist of exercises for the upper and lower limbs. Initially, the patients will perform 2 sets of 10 repetitions with load of 50% to 70% of 1-RM and the progression will take place in the number of repetition, and then in the load.
  Arms: Exercise, dietary and behavioral therapy
Other: Stretching and Breathing exercise — Breathing exercise will consist of 3 exercises adapted from yoga's breathing technique (kapalabhati, uddhiyana and agnisara) twice a week, totaling 24 sessions of 30 minutes each. Every exercise will be performed in sets of 3 (2 minutes each) with 60 seconds of rest between them. The stretching will consist of stretching exercises for the major muscle groups in 3 sets of 10 seconds each. The program will be performed twice a week, totaling 24 sessions of 30 minutes each.
  *Both breathing and stretching exercises will be performed as placebo to ensure the same duration of treatment between the two groups.
  Arms: Dietary and behavioral therapy

SUMMARY:
Obese asthmatics have more severe symptoms, reduced lung function, poorer quality of life and a reduced response to inhaled corticosteroid medication compared to non-obese asthmatics. In addition, the impact of a weight-loss program on clinical control and psychological outcomes has been poorly demonstrated and the effect of exercise training remain unknown. The investigators aim to investigate the effect of exercise training in a weight-loss program on asthma clinical control (primary outcome), health factors related to quality of life and psychosocial symptoms (secondary outcomes) in obese patients with moderate-to-severe persistent asthma. Physical activity, inflammatory profiles and sleep disorders will also be evaluated. The investigators' hypothesis is that exercise as part of a weight-loss program is more effective to lose weight and improve asthma control, quality of life and psychosocial symptoms in obese asthmatics.

DETAILED DESCRIPTION:
This is a randomized, controlled and single blinded trial. Fifty-four asthmatic adults will be randomly assigned into two groups: DBG (dietary and behavioral support group) or DBE (similar to DBG + exercise training). Both groups will complete a weight-loss program based on dietary and behavioral therapy. In addition, DBE will perform a training program based on aerobic and resistance training whereas DBG will perform a breathing and stretching program. Interventions will be performed twice a week for 3 months, 60 minutes each. The data normality will be analyzed by Kolmogorov-Smirnov, the variables obtained before interventions will be compared with the Student t-test or Mann-whitney U-test. Comparisons of the initial and final data on outcomes will be analyzed with repeated measures ANOVA with appropriate post hoc of Bonferroni. The significance level will be set to 5% for all tests.

ELIGIBILITY:
Inclusion Criteria:

* Asthma moderate and severe
* Asthma will diagnosed (Global Initiative for Asthma -GINA)
* Body Mass Index between 35 kg/ m2 and 39,9 kg/m2
* Sedentary
* Medical treatment, for at least 6 months
* Clinically stable (i.e., no exacerbation or medication changes for at least 30 days)

Exclusion Criteria:

* Cardiovascular, musculoskeletal or other chronic lung diseases
* Active Cancer
* Pregnant
* Weight loss more than 5 % in the preceding 6 months
* Using weight-loss medications
* History of bariatric surgery, uncontrolled hypertension or diabetes
* Using overnight continuous positive airway pressure
* Lactating
* Current or ex-smoker

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2014-07; Primary Completion 2015-02 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Clinical Control | Before and after 3 months of intervention
  Clinical control will be evaluated by asthma control questionnaire (ACQ)

SECONDARY OUTCOMES:
Health related quality of life | Before and after 3 months of intervention
  Health related quality of life will be assessed by Asthma Quality Life Questionnaire (AQLQ)
Level of depression and anxiety | Before and after 3 months of intervention
  the symptoms of depression and anxiety will be assessed by Hospital Anxiety and Depression (HAD)

OTHER OUTCOMES:
Airway inflammation | Before and after 3 months of intervention
  Airway inflammation will be quantified using the exhaled fraction of nitric oxide (FeNO)
serum cytokines and adipokines levels | Before and after 3 months of intervention
  The method Cytometric Beat Array (CBA) (BD Biosciences, USA) will be used to analyze the levels of interleukins (IL) IL-4, IL-5, IL-6, IL-8, IL -10,IL-1ra, IL-13,Tumor Necrosis Factor (TNF-α), leptin, adiponectin and C-reactive protein (CRP)
Daily life physical activity | Before and after 3 months of intervention
  Daily life physical activity will be assessed using an accelerometer (actigraph activity monitor) and physical capacity will be assessed by an incremental cardiopulmonary exercise testing
Sleep disorders | Before and after 3 months of intervention
  sleep disorders will be assessed by Berlin Questionnaire for Sleep Apnea and Actisleep activity monitor
Lung function | Before and after 3 months of intervention
  Static and dynamic lung volumes will be assessed by Spirometry and Plethysmograph
Physical fitness | Before and after 3 months of intervention
  Aerobic potency will be assessed by Cardiopulmonary exercise test
Asthma symptoms and exacerbations | Before and after 3 months of intervention
  Asthma symptoms will be assessed using a daily diary of symptoms and exacerbation will be defined by an increase in symptoms associated with at least one of the following criteria: use of rescue medication ≥4 puffs per 24 hours during a 48-hour period, need for systemic corticosteroids, unscheduled medical appointment, visit to an emergency room or hospitalization.
Body composition | Before and after 3 months of intervention
  Body composition will be analyzed by using a tetrapolar 8-point tactile bioelectrical impedance

CONTACTS AND LOCATIONS:
Overall Officials: Celso RF Carvalho, PhD, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- Clinical Hospital of São Paulo University medical school (HCFMUSP), São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Freitas PD, Ferreira PG, Silva AG, Stelmach R, Carvalho-Pinto RM, Fernandes FL, Mancini MC, Sato MN, Martins MA, Carvalho CR. The Role of Exercise in a Weight-Loss Program on Clinical Control in Obese Adults with Asthma. A Randomized Controlled Trial. Am J Respir Crit Care Med. 2017 Jan 1;195(1):32-42. doi: 10.1164/rccm.201603-0446OC. PMID 27744739
- [Derived] Freitas PD, Ferreira PG, da Silva A, Trecco S, Stelmach R, Cukier A, Carvalho-Pinto R, Salge JM, Fernandes FL, Mancini MC, Martins MA, Carvalho CR. The effects of exercise training in a weight loss lifestyle intervention on asthma control, quality of life and psychosocial symptoms in adult obese asthmatics: protocol of a randomized controlled trial. BMC Pulm Med. 2015 Oct 21;15:124. doi: 10.1186/s12890-015-0111-2. PMID 26487563